CLINICAL TRIAL: NCT05381909
Title: A Phase 1 Study Investigating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Antitumor Activity of Second Mitochondrial-derived Activator of Caspases Mimetic BGB-24714 as Monotherapy and With Combination Therapies in Patients With Solid Tumors
Brief Title: A Study of BGB-24714 as Monotherapy and With Combination Therapies in Participants With Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The research was terminated voluntarily due to changes in the company's business strategy regarding the development of BGB-24714, rather than any safety issues.
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-24714-101; CTR20232532 (Other: ChinaDrugTrials)
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumor, Adult
Keywords: Solid tumors; Advanced Solid Tumors; Metastatic Solid Tumors
MeSH Terms: interventions — Paclitaxel; Carboplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Phase 1a: Dose Escalation Part A (Experimental): Participants will receive escalating doses of BGB-24714 as monotherapy
  Interventions: Drug: BGB-24714
- Phase 1a: Dose Escalation Part B (Experimental): Participants will receive increasing dose levels of BGB-24714 in combination with paclitaxel
  Interventions: Drug: BGB-24714; Drug: Paclitaxel
- Phase 1a: Dose Escalation Part C (Experimental): Participants will receive increasing dose levels of BGB-24714 in combination with chemoradiation
  Interventions: Drug: BGB-24714; Drug: Paclitaxel; Drug: Carboplatin
- Phase 1a: Dose Escalation Part D (Experimental): Participants will receive increasing dose levels of BGB-24714 in combination with chemoradiation
  Interventions: Drug: BGB-24714; Drug: Paclitaxel; Drug: Carboplatin
- Phase 1a: Dose Escalation Part A-CN (Experimental): Participants will receive escalating doses of BGB-24714 as monotherapy in Chinese participants
  Interventions: Drug: BGB-24714
- Phase 1a: Dose Escalation Part E (Experimental): Participants will receive increasing dose levels of BGB-24714 in combination with chemoradiation in Chinese participants
  Interventions: Drug: BGB-24714; Drug: Paclitaxel; Drug: Carboplatin
- Phase 1b: Dose Expansion (Experimental): BGB 24714 will be administered in combination with paclitaxel or docetaxel in participants with selected solid tumors.
  Interventions: Drug: BGB-24714; Drug: Paclitaxel; Drug: Docetaxel

INTERVENTIONS:
Drug: BGB-24714 — administered orally
Drug: Paclitaxel — administered intravenously
  Arms: Phase 1a: Dose Escalation Part B; Phase 1a: Dose Escalation Part C; Phase 1a: Dose Escalation Part D; Phase 1a: Dose Escalation Part E; Phase 1b: Dose Expansion
Drug: Carboplatin — administered intravenously
  Arms: Phase 1a: Dose Escalation Part C; Phase 1a: Dose Escalation Part D; Phase 1a: Dose Escalation Part E
Drug: Docetaxel — administered intravenously
  Arms: Phase 1b: Dose Expansion

SUMMARY:
This study aims to understand how safe and well-tolerated a drug called BGB-24714 is when used alone, or in combination with chemotherapy or radiation therapy, for people with advanced or spreading solid tumors. The main objective is to identify the highest tolerable dose or the highest administered dose of BGB-24714. Additionally, the study aims to identify the most suitable doses for further investigation in larger groups of participants.

ELIGIBILITY:
Key Eligibility Criteria :

1. Participants must sign a written informed consent form (ICF); and agree to comply with study requirement
2. Phase 1a (Dose Escalation):

   Part A, A-CN, and B: Participants with histologically or cytologically confirmed unresectable locally advanced or metastatic solid tumor previously treated with standard systemic therapy or for whom treatment is not available or not tolerated Note: Only Chinese participants will be eligible for Part A-CN.

   Part C: Participant has histologically or cytologically confirmed, locally advanced, unresectable Stage III Non-small cell lung cancer (NSCLC) suitable for definitive chemoradiotherapy (CRT)

   Part D: Participant with locally advanced, histologically confirmed inoperable esophageal squamous cell carcinoma (ESCC) suitable for definitive CRT

   Phase 1b (Dose Expansion): Participants with histologically or cytologically confirmed solid tumors of selected types previously treated with standard therapy.
3. Participants must be able to provide formalin-fixed paraffin embedded (FFPE) tumor tissue sample.
4. Phase 1a Part A, A-CN, B and Phase 1b: ≥ 1 measurable lesion per Response evaluation criteria in solid tumors (RECIST) v1.1
5. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1

Key Exclusion Criteria:

1. Active leptomeningeal disease or uncontrolled, untreated brain metastasis.
2. Any malignancy ≤ 3 years before the first dose of study drug(s) except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated with curative intent
3. Any condition that required systemic treatment with either corticosteroids or other immunosuppressive medication ≤ 14 days before the first dose of study drug(s).
4. Clinically significant infection requiring systemic therapy ≤ 14 days before the first dose of study drug(s).
5. Prior exposure to agents with second mitochondria-derived activator of caspases (SMAC) mimetics, or other Inhibitors of apoptosis proteins (IAPs) antagonists.

NOTE: Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Dose Escalation: Number of participants with adverse events (AEs) | approximately 6 months
  Number of participants with treatment-emergent adverse events (TEAEs), serious adverse events (SAEs ), and experiencing AEs meeting protocol defined Dose-Limiting Toxicity (DLT) criteria.
Dose Escalation: Maximum tolerated dose (MTD) of BGB-24714 as monotherapy, in combination with chemotherapy, and in combination with concurrent chemoradiotherapy (cCRT) | approximately 6 months
Dose Escalation: Recommended Doses for Expansion (RDFE) of BGB-24714 as monotherapy, in combination with chemotherapy, and in combination with concurrent chemoradiotherapy (cCRT) | approximately 6 months
  Recommended dose based upon the MTD or MAD, as well as the long-term tolerability, pharmacokinetics, efficacy, and any other relevant data as available
Dose Expansion: Objective response rate (ORR) | approximately 2 Years
  ORR is defined as the percentage of participants with partial or complete response, as determined by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)

SECONDARY OUTCOMES:
Dose Escalation: Objective response rate (ORR) | approximately 2 Years
  ORR is defined as the percentage of participants with partial or complete response, as determined by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Dose Expansion: Progression-free Survival (PFS) | approximately 2 Years
  PFS is defined as the time from the date of the first dose of study drug to the date of first documentation of disease progression as determined by the investigator using RECIST v1.1 or death, whichever occurs first
Dose Expansion: Number of participants with adverse events | approximately 2 Years
  Number of participants with AEs and SAEs
Duration of Response (DOR) | approximately 2 Years
  DOR is defined as the time from the date that response criteria are first met to the date that progressive disease is objectively documented or death, whichever comes first as determined by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Disease Control Rate (DCR) | approximately 2 Years
  DCR is defined as the percentage of participants whose best overall response is complete response, partial response, or stable disease, as determined by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Clinical Benefit Rate (CBR) | approximately 2 Years
  CBR is defined as the percentage of participants who have complete response, partial response, and stable disease, as determined by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Plasma Concentrations of BGB-24714 and its metabolite | approximately 2 Years
Maximum Observed Plasma Concentration (Cmax) of BGB-24714 and its metabolite | Up to 48 hours postdose
Time to Maximum Plasma Concentration (Tmax) of BGB-24714 and its metabolite | Up to 48 hours postdose
Terminal Half-life (t1/2) of BGB-24714 and its metabolite | Up to 48 hours postdose
Area Under the Plasma Concentration Time Curve from Time 0 to the Last Quantifiable Concentration (AUC0-last) of BGB-24714 and its metabolite | Up to 48 hours postdose
Area Under The Plasma Concentration Time Curve From Time 0 To Infinity (AUC0-inf) of BGB-24714 and its metabolite | Up to 48 hours postdose
Apparent Clearance (CL/F) of BGB-24714 | Up to 48 hours postdose
Apparent Volume Of Distribution (Vz/F) of BGB-24714 | Up to 48 hours postdose
Concentration at steady state (Cmax,ss) of BGB-24714 and its metabolite | Up to 48 hours postdose
Time to Maximum Plasma Concentration at steady state (Tmax,ss) of BGB-24714 and its metabolite | Up to 48 hours postdose
Area Under the Plasma Concentration Time Curve from Time 0 to the Last Quantifiable Concentration at Steady State (AUClast,ss) of BGB-24714 and its metabolite | Up to 48 hours postdose
Rough Concentration At Steady State (Ctrough,ss) of BGB-24714 and its metabolite | Up to 48 hours postdose

CONTACTS AND LOCATIONS:
Locations (34):
- United States (17):
  - Banner Md Anderson Cancer Center, Gilbert, Arizona
  - Florida Cancer Specialist (Scri) Sarasota, Sarasota, Florida
  - Scri Florida Cancer Specialists North, St. Petersburg, Florida
  - Scri Florida Cancer Specialist East, West Palm Beach, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Upmc Hillman Cancer Center(Univ of Pittsburgh), Pittsburgh, Pennsylvania
  - Sanford Cancer Center, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Tennessee Oncology, Pllc Nashville, Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The University of Texas Md Anderson Cancer Center (Department Gi Medical Oncology), Houston, Texas
  - Intermountain Healthcare, Salt Lake City, Utah
  - Next Virginia, Fairfax, Virginia
  - University of Washington, Seattle, Washington
- Australia (6):
  - Northern Beaches Hospital, Frenchs Forest, New South Wales
  - Icon Cancer Centre South Brisbane, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Austin Health, Heidelberg, Victoria
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
  - Sunshine Hospital, St Albans, Victoria
- China (5):
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Shandong Provincial Hospital, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
- Auckland City Hospital, Auckland, New Zealand
- South Korea (5):
  - National Cancer Center (Korea), IlsandongGu GoyangSi, Gyeonggi-do
  - Gachon University Gil Medical Center, NamdongGu, Incheon Gwang'yeogsi
  - Samsung Medical Center, GangnamGu, Seoul Teugbyeolsi
  - Severance Hospital Yonsei University Health System, SeodaemunGu, Seoul Teugbyeolsi
  - Asan Medical Center, SongpaGu, Seoul Teugbyeolsi

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/